CLINICAL TRIAL: NCT03519438
Title: Evaluating the Efficacy of Mepitel in Post-mastectomy Breast Cancer Patients, and Examining the Role of the Skin Microbiome in Radiation Dermatitis
Brief Title: Evaluating Mepitel in Post-mastectomy Patients and the Role of the Skin Microbiome in Radiation Dermatitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kimberly S. Corbin, Assistant Professor, Radiation Oncology, Mayo Clinic
Other Study IDs: 17-001546; ROR1701 (Other: Mayo Clinic)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — mepitel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Lateral 3/4 of treatment field: placement of Mepitel on the lateral ¾ of the treatment field
  Interventions: Other: Mepitel
- Medial 3/4 of treatment field: placement of Mepitel on the medial ¾ of the treatment field
  Interventions: Other: Mepitel

INTERVENTIONS:
Other: Mepitel — Mepitel film will be placed on 3/4 of treatment field to protect from radiation dermatitis

SUMMARY:
The aim of this study is to examine alterations in the skin microbiome that occur during radiation therapy. The study design will examine changes secondary to ionizing radiation, and correlate these changes with the development and severity of radiation dermatitis. The goal is to improve understanding of the mechanism of radiation dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histological confirmation of breast or chest wall malignancy
* Primary or recurrent disease eligible
* Post-mastectomy with or without reconstruction
* Undergoing unilateral external beam radiotherapy at the Mayo Clinic - Rochester, MN or Mayo Clinic - Eau Claire, WI
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to consent for photography of radiation field
* Available to return to Mayo Clinic in within 6 weeks post-treatment for assessment
* Able to initiate thin film usage within first 3 days of the initiation of treatment

Exclusion Criteria:

* Documented history of adhesive or tape allergy
* Unable to provide written consent
* Patients with prior radiotherapy to any portion of the planned treatment site
* Brachytherapy patients
* Patients with active rash, pre-existing dermatitis, lupus, or scleroderma
* Gross dermal involvement at initiation of radiotherapy
* Recent use of systemic or topical antibiotics or antifungal medications within 14 days of swab collection
* Recent use of any of the following within 14 days of swab collection:

  * Systemic or topical steroids
  * Use of systemic immunosuppressant drugs
  * Use of ultraviolet light therapy
* Clinical evidence of infection that in the judgement of the principle investigator would interfere with proper assessment of the skin microbiome
* Prior organ or bone marrow transplant
* Current lactation
* Undergoing bilateral radiation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: post-mastectomy breast cancer patients
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
severity of radiation dermatitis in irradiated skin protected by Mepitel Film dressing versus uncovered skin receiving standard skin treatment | 12 weeks
changes in the skin microbiome that occur secondary to ionizing radiation including quantitative analysis of S. aureus | 12 weeks
changes in the skin microbiome of patients who use Mepitel including quantitative analysis of S. aureus | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Corbin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials